CLINICAL TRIAL: NCT03971864
Title: The Relationship Between Peripheral Artery Plaque Characteristics Evaluated by Ultrasound and Coronary Culprit Lesion Characteristics Evaluated by OCT in ACS Patients
Brief Title: Peripheral Vascular Disease and Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director of Cardiology of The Seconf Affiliated Hospital of Harbin Mdical University, Harbin Medical University
Other Study IDs: HMUOCT-PAU
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at evaluating the relationship between peripheral artery plaque characteristics evaluated by ultrasound and coronary culprit lesion characteristics evaluated by OCT in ACS patients.

DETAILED DESCRIPTION:
Patients with acute coronary syndrome (ACS) who underwent percutaneous coronary intervention (PCI) and optical coherence tomography (OCT) are included in this study. Two skillful echocardiographers will evaluate peripheral artery plaque characteristics by ultrasound.Ultrasound parameters of peripheral artery will be compared among patients with different coronary culprit lesion characteristics, such as plaque rupture and plaque erosion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as ACS underwent coronary angiography and OCT examination
* Agreed to accept peripheral artery ultrasound examination

Exclusion Criteria:

* In-stent restenosis, coronary dissection, coronary spam, thrombus
* left main artery disease
* Age>85 years old
* Cardiogenic shock or stroke admission
* Severe hepatic or renal dysfunction
* Poor quality of OCT image or massive thrombus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS patients
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Differences in ultrasound parameters of peripheral artery plaque according to different coronary culprit lesion morphology. | Baseline
  Plaque rupture is characterized by the presence of fibrous cap discontinuity with a cavity formation. plaque erosion is characterized by the presence of the attached thrombus overlying an intact and visual plaque, luminal surface irregularity at the culprit lesion in the absence of thrombus, or attenuation of the underlying plaque by thrombus without superficial lipid or calcification immediately proximal or distal to the site of thrombus.Patients with plaque erosion have less plaques, lower intima-media thickness (IMT), lower plaque score (PS) compared to patients with plaque rupture.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weng Z, Zhao C, Qin Y, Liu C, Pan W, Hu S, He L, Xu Y, Zeng M, Feng X, Gao R, Yu X, Liu M, Yi B, Zhang D, Koniaeva E, Musin T, Mohammad D, Zhu B, Sun Y, Hou J, Tian J, Mintz GS, Jia H, Yu B. Peripheral atherosclerosis in acute coronary syndrome patients with plaque rupture vs plaque erosion: A prospective coronary optical coherence tomography and peripheral ultrasound study. Am Heart J. 2023 Sep;263:159-168. doi: 10.1016/j.ahj.2023.06.006. Epub 2023 Jun 14. PMID 37327980